CLINICAL TRIAL: NCT05395494
Title: A Randomized Controlled Trial of Adjunctive D-Cycloserine to Intermittent Theta-burst Stimulation Transcranial Magnetic Stimulation in Fibromyalgia
Brief Title: iTBS-DCS in Fibromyalgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility criteria met on interim analysis
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB21-1916
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- D-Cycloserine (Experimental): Participants will orally ingest a capsule containing 100mg of the antibiotic d-cycloserine daily (Monday-Friday) during 4 weeks of rTMS treatment (20 sessions) 60-120 minutes prior to rTMS treatment.
  Interventions: Drug: D-Cycloserine; Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS)
- Placebo (Placebo Comparator): Participants will orally ingest a capsule identical to that containing the study medication, however this capsule will contain a placebo. They will ingest this capsule daily (Monday-Friday) for 4 weeks of rTMS treatment (20 sessions) 60 - 120 minutes prior to rTMS treatment.
  Interventions: Drug: Placebo oral tablet; Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Drug: D-Cycloserine — Daily oral D-cycloserine 100mg during TMS treatments (20 days).
  Other Names:
  Seromycin
  Other Names: Seromycin
  Arms: D-Cycloserine
Drug: Placebo oral tablet — Daily oral placebo during the TMS treatments (20 days).
  Arms: Placebo
Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS) — Repetitive Transcranial magnetic stimulation (rTMS) will be delivered using a MagPro X100 device with B70 coil and the intermittent theta burst (iTBS) protocol to the left dorsolateral prefrontal cortex. Participants will receive daily treatments (Monday-Friday) over four weeks.

SUMMARY:
Background & Rationale: Fibromyalgia is characterized by widespread pain, fatigue, mood and anxiety as well as cognitive complaints. For an unacceptable proportion of patients, depressive symptoms remain impairing despite multiple treatments.

For such patients, novel treatments include non-invasive brain stimulation. Transcranial Magnetic Stimulation (TMS) targeting the dorsolateral prefrontal cortex (DLPFC) or the primary motor cortex (M1) is the non-invasive neurostimulation method with the largest evidence base in fibromyalgia. It involves generating magnetic fields outside of the body to change the firing of neurons in the brain, and has a very favorable tolerability profile. Recent meta-analyses indicate that both the DLPFC and M1 targets are associated with improvements in pain, mood and anxiety, however the benefits are more persistent when the DLPFC is targeted (Su et al, 2021 - J Clin Med). The DLPFC is important in fibromyalgia through its implication in several symptoms domains in fibromyalgia, as well as pain catastrophization.

The researchers neurophysiological data and clinical data in depression suggests that the researchers can enhance the effects of TMS by using an adjunctive medication called D-Cycloserine (DCS, 100mg) in conjunction with a protocol called intermittent theta-burst stimulation (iTBS). Specifically, this data indicated that several converging features of fibromyalgia improve with augmented iTBS, specifically depressive symptoms, anxiety symptoms, fatigue, and cognitive function. The researchers therefore hypothesize that the combination of D-cycloserine and TMS will lead to greater improvements in fibromyalgia symptoms than TMS alone.

Although iTBS has not yet been studied in fibromyalgia, it has a well characterized neurophysiological effect and been shown to be non-inferior to conventional TMS protocols in conditions such as depression. More importantly, its physiological basis can be manipulated with D-Cycloserine whereas this has not been convincingly demonstrated with rTMS (see Brown et al, 2019, 2021 Brain Stim).

Research Question and Objectives: To conduct a randomized placebo-controlled trial of DCS in adjunct with rTMS in Fibromyalgia. Participants will be randomized to receive 100mg of DCS or placebo together with TMS.

DETAILED DESCRIPTION:
Methods: 90participants (males and females aged aged 18-65, with a diagnosis of fibromyalgia of at least moderate moderate impact as defined by a FIQR score of ≥39, stable psychotropic medication for 4 weeks) will be recruited. Patients will be randomized 1:1 to TMS+DCS or TMS+Placebo. Participants who do not have recent bloodwork will have laboratory tests to rule out haematological, hepatic, and renal disease, and participants will be screened for suicidal ideation. The dose of DCS will be 100mg, taken daily for four weeks. Clinical outcomes will be quantified using the Revised Fibromyalgia Impact Questionnaire (FIQR), as well as clinical and self reported measures of depression, anxiety, and quality of life done at baseline, halfway through TMS treatment (week 2), and after TMS treatment (week 4). Participants clinical symptoms will be evaluated again one-month after treatment (week 8). Quantitative sensory testing done at baseline and week 4 will characterize sensory perception. Blood samples at baseline and week 4 will be used to analyze changes in pro-inflammatory markers. Changes in cognition will be assessed by cognitive testing at baseline, week 4, and week 8. MRI scans completed at baseline and week 4. MRI scans at baseline and week 4 will be used to assess the following neuroimaging outcomes: single voxel magnetic resonance spectroscopy, locus coeruleus neuromelanin, and functional MRI resting state connectivity.

In parallel, a matched sample of 90 healthy participants will be cross-sectionally characterized for normative comparison, and these participants will not go on to receive any TMS or other interventions. Having this sample of healthy participants will allow the researchers to determine the clinical, cognitive, sensory, and imaging characteristics that characterize fibromyalgia. They will also allow the researchers to determine whether treatment effects restore clinical, cognitive, sensory, and imaging characteristics to the level of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 65 years
2. are competent to consent to treatment
3. have a diagnosis of fibromyalgia as per the American College of Rheumatology 2016 fibromyalgia criteria.
4. have failed to achieve a clinical response to an adequate trial of a serotonin reuptake inhibitor, a norepinephrine reuptake inhibitor, cognitive behavioral therapy or have been unable to tolerate these medications/access psychotherapy.
5. have a score ≥ 41 on the FIQR.
6. have had no change in dose, or initiation of any psychotropic medication in the 4 weeks prior to randomization
7. are able to adhere to the treatment schedule
8. pass the TMS adult safety screening (TASS) and MRI screening questionnaire
9. have had blood work within the last month (complete blood count, electrolytes, BUN, creatinine, eGFR, AST, ALT and GGT) within the reference range.

Exclusion Criteria:

1. Allergy to cycloserine or any excipients.
2. have an alcohol or substance use disorder within the last 3 months
3. have suicidal ideation (score of 4 ≥ on item 10 of MADRS or positive response to item 4 on the CSSRS-screen)
4. are at a significant risk of harm to themselves or others
5. current symptoms of psychosis
6. history of psychosis
7. are currently pregnant, breast feeding or plan to become pregnant. Health Canada requires that women of reproductive potential utilize either highly effective birth control or double barrier method of contraception. Abstinence is only acceptable when it is the usual and preferred lifestyle of the participant.
8. history of non-response to rTMS treatment.
9. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of epilepsy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
10. have concomitant major unstable medical illness, cardiac pacemaker, or implanted medication pump
11. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
12. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
13. are currently (or in the last 4 weeks) not taking any benzodiazepine, cyclopyrrolone, gabapentin/pregabalin or anticonvulsant due to the potential to limit iTBS efficacy
14. are being currently treated with ethionamide or isoniazid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Change in severity of the impact of fibromyalgia as measured by the Revised Fibromyalgia Impact Questionnaire (FIQR). The FIQR is a self-administered questionnaire commonly used to evaluate fibromyalgia across 3 domains: function, overall impact and symptoms. The FIQR consists of 21 individual questions, each with a rating scale of 0 (no impact) -10 (maximum impact).
Sustained changes in Revised Fibromyalgia Impact Questionnaire (FIQR) | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Differences in sustained treatment effects between iTBS+cycloserine and iTBS+placebo groups as measured by Revised Fibromyalgia Impact Questionnaire (FIQR) changes one month after treatment end. The FIQR is a self-administered questionnaire commonly used to evaluate fibromyalgia across 3 domains: function, overall impact and symptoms. The FIQR consists of 21 individual questions, each with a rating scale of 0 (no impact) -10 (maximum impact).
Differential change in the primary outcome will be mediated by D-Cycloserine plasma level | Single timepoint. First day of TMS treatment, 90 minutes after ingestion of blinded oral capsule.
  Participants will provide a blood sample prior to the first TMS treatment (90 minutes after ingestion of blinded oral capsule) to characterize D-Cycloserine plasma levels. The primary efficacy measures will be examined in relation to drug blood levels.
Differential change in the primary outcome will be mediated by fidelity to the protocol | Daily Monday-Friday throughout study (4 weeks)
  All participants will be instructed to take the blinded capsule 60 - 120 minutes prior to TMS treatment, ensuring adequate time for drug absorption. Daily logs will be kept by the study staff to confirm time of capsule ingestion and TMS treatment. Any TMS sessions missed, capsule doses missed and/or capsule doses taken at the incorrect time will be tracked. The primary efficacy measures will be examined in relation to adherence to the protocol (20/20 TMS session completed with oral capsule taken between 60 - 120 minutes prior).

SECONDARY OUTCOMES:
Change in Physical Function as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  Domain 1 assesses physical function through 4 questions scored from 1-5, with lower scores indicating greater impairment. Suggested interpretation of total scores below:
  15- 20 = Acceptable/ mild 7 - 15 = Moderate concern 4 - 6 = Significant concern
Change in Anxiety as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  Domain 2 assesses anxiety through 4 questions scored from 1-5, with higher scores indicating greater levels of anxiety. Suggested interpretation of total scores below:
  4-10 = Acceptable/ mild 11-15 = Moderate concern 16-20 = Significant concern
Change in Depression as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  Domain 3 assesses depression through 4 questions scored from 1-5, with higher scores indicating increased depressive symptoms. Suggested interpretation of total scores below:
  4-10 = Acceptable/ mild 11-16 = Moderate concern 17-20 = Significant concern
Change in Fatigue as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  Domain 4 assesses Fatigue through 4 questions scored from 1-5, with higher scores indicating greater fatigue. Suggested interpretation of total scores below:
  4-13 = Acceptable/ mild 14-18 = Moderate concern 19-20 = Significant concern
Change in Sleep Disturbances as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  Domain 5 assesses sleep quality through 4 questions scored from 1-5, with higher scores indicating greater sleep disturbances. Suggested interpretation of total scores below:
  4-15 = Acceptable/ mild 16-19 = Moderate concern 20 = Significant concern
Change in Social Function as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  Domain 6 assesses ability to participate in social roles/activities through 4 questions scored from 1-5, with lower scores indicating greater impairment. Suggested interpretation of total scores below:
  10- 20 = Acceptable/ mild 5 - 9 = Moderate concern 4 = Significant concern
Change in Pain Interference as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  Domain 7 assesses pain interference through 4 questions scored from 1-5, with higher scores indicating higher pain interference. Suggested interpretation of total scores below:
  4 -11 = Acceptable/ mild 12-18 = Moderate concern 19-20 = Significant concern
Change in Pain Intensity as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS-29 is a 29 item questionnaire that assesses 7 domains: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, pain interference, and a 0-10 pain intensity scale.
  The Pain intensity scale asks individuals to rate their pain on a scale from 0 to 10, where 0 is no pain and 10 is the worst possible pain.
Change in self-reported pain as measured by the Short-Form McGill Pain Questionnaire (SF-MPQ) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Short-Form McGill Pain Questionnaire (SF-MPQ) is a self-reported measurement of pain consisting of 15 descriptive items and two overall pain scales. The descriptive items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. The scale for present pain intensity is rated from 0 (no pain) to 5 (excruciating pain) and a average pain intensity is rated on a 10-point visual analogue scale (VAS), with 0 representing no pain and 10 representing the worst possible pain.
  The measure is calculated by summing the point values for responses to 15 questions and the two scales, with totals ranging from 0 (no pain) to 60 (worst possible pain).
Change in self-reported pain as measured by the painDETECT scale. | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  painDETECT is a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain. A total score that ranges from -1 to 38 can be calculated from the nine items, with higher scores indicating higher levels of pain.
Change in Central Sensitization Pain as measured by the The Central Sensitization Inventory (CSI) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Central Sensitization Inventory (CSI) is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitivity syndromes such as fibromyalgia, neck injury, temporomandibular joint disorder or migraine/tension headaches. The CSI may be used to determine severity of chronic centralized pain. The CSI consists of 25 questions and may be self-administered. Each question may be answered as follows: Never(0points), Rarely(1point), Sometimes(2points), Often(3points), or Always(4points). Total points reflect the severity of the central sensitization pain.
  Following is a break down of score ranges and the intensity of central sensitization pain they represent.
  Subclinical: 0 to 29 Mild: 30 to 39 Moderate: 40 to 49 Severe: 50 to 59 Extreme: 60 to 100
Change in fibromyalgia severity as measured by the Polysymptomatic Distress Scale (PDS). | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The polysymptomatic distress scale (PDS) provides an overall measure of pain extent and symptom distress, and is considered a measure of fibromyalgia severity. The scale total ranges from 0 to 31, with higher scores indicating greater severity.
Montgomery-Asberg Depression Rating Scale (MADRS) | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Change in severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Number of participants with clinical depression remission | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Clinical remission of depressive symptoms will be measured by the Montgomery-Asberg Depression Rating Scale (MADRS); a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. A score of </= 10 on the MADRS indicates clinical remission.
Number of participants with clinical depression response | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Clinical depression response will be measured by the Montgomery-Asberg Depression Rating Scale (MADRS); a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. A reduction of >/= 50% in the MADRS score indicates clinical response.
Clinical Global Impression- Severity | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The CGI-Severity scale is clinician rated from 1-7 representing 'Not at all ill' to 'Severely ill'.
Clinical Global Impression- Improvement | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The CGI-Improvement scale is a clinician rated 1-7, representing the range between 'Very much improved' and 'Very much worse' from the baseline visit.
Changes in self-reported depression as measured by the Quick Inventory of Depressive Symptoms (QIDS-SR) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Quick Inventory of Depressive Symptomatology (QIDS) rates depression symptoms via self-assessment.Severity of depression can be judged based on the total score.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
Changes in self-reported anxiety as measured by the Generalized Anxiety Disorder (GAD-7) questionnaire | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Anxiety symptoms will be assessed using the 7 item Generalized Anxiety Disorder (GAD-7) questionnaire. The GAD-7 measures self-reported feelings of anxiety within the last 2 weeks. Scores range from 0-21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
Changes in self-reported depression and anxiety as measured by the The Hospital Anxiety and Depression Scale (HADS) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Hospital Anxiety and Depression Scale (HADS) is a self-rating scale developed to assess psychological distress in non-psychiatric patients. It consists of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression. The total score is the sum of the 14 items. A higher score indicates higher distress.
Changes in sleep quality as measured by the The Insomnia Severity Index (ISI) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Insomnia Severity Index (ISI) is a brief, 7 question instrument that was designed to assess the severity and symptoms of insomnia. The seven answers are added up to get a total score, with higher scores indicating greater severity of insomnia.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Changes in general health as measured by a visual analog scale (VAS) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  A Visual Analog Scale (VAS) will ask participants how good or bad their overall health is today. This scale is numbered from 0 to 100. 100 indicates the best health they can imagine. 0 indicates the worst health they can imagine.
Change in quality of Life as measured by the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The WHOQOL-BREF is a self-reported questionnaire which assesses individual's perception of their quality of life across 4 domains; physical health, psychological, social relationships and environment. Domains scores are calculated to range from 0-20 and scaled in a positive direction (ie. higher scores denote higher quality of life).
Change in fatigue symptoms as measured by the Chalder Fatigue Questionnaire | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Chalder Fatigue Questionnaire is an 11-item questionnaire measuring the severity of physical and mental fatigue. Each question uses a 4-point Likert scale with higher values representing greater symptoms. The respondent's global score can range from 0 (no symptoms) to 33 (most symptomatic). The global score can be further split into two dimensions-physical fatigue (measured by items 1-7) and psychological fatigue (measured by items 8-11).
Changes in catastrophic thinking related to pain using the Pain Catastrophizing Questionnaire (PCQ) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Pain Catastrophizing Questionnaire (PCQ) is a 13-item instrument for measuring catastrophic thinking related to pain. People are asked to indicate the degree to which they have catastrophizing thoughts and feelings when they are experiencing pain on 5-point Likert scales, from (0) note at all to (4) all the time.
  A total score is yielded (ranging from 0-52), with higher scores indicating higher levels of catastrophizing. The total score can further be split into three subscale scores, assessing rumination (sum of items 8, 9, 10 and 11. Range of 0-16), magnification (sum of items 6, 7, and 13. Range of 0-12), and helplessness (sum of items 1, 2, 3, 4, 5, and 12. Range of 0-24).
  Total scores of above 30 indicates clinically relevant level of catastrophizing.
Change in self-reported personality traits as measured by the Big Five Inventory (BFI) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Big Five Inventory (BFI) is a self-report inventory designed to measure the Big Five dimensions of personality: extroversion, agreeableness, openness, conscientiousness, and neuroticism. The test consists of 44 items that you must rate on how true they are about you on a five point scale where 1=Disagree, 3=Neutral and 5=Agree.
Changes in pain medication usage | Data will be collected at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Participants will be asked to list all medications they have used in the last week to manage pain, including prescription and over the counter treatments.
Change in self reported cognitive failures as measured by The Cognitive Failures Questionnaire (CFQ) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Cognitive Failures Questionnaire (CFQ) is used to assess the frequency with which people experienced cognitive failures, such as absent-mindedness, in everyday life -- slips and errors of perception, memory, and motor functioning.
  Individuals are asked to rate how often they experience different cognitive failures from "never "(0) to "very often" (4). The sum of the ratings of the 25 individual items yields a score from 0-100, with higher scores indicating more cognitive failures.
Change in self reported cognitive function as measured by The Multidimensional Inventory of Subjective Cognitive Impairment (MISCI) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The Multidimensional Inventory of Subjective Cognitive Impairment is a 10-item instrument to evaluate subjective cognitive function in patients with fibromyalgia. Each item consists of a statement regarding cognitive abilities in the past week and responders are asked to agree with each statement on a 5-point Likert scale, from 1 (not at all/never) to 5 (very much/always).
  Scoring: 4 negatively-worded items (item 7 - 10) from the MISCI are reverse scored. Items are summed to receive a total score ranging from 10 to 50, with higher total scores indicative of better subjective cognitive functioning.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Perceived Deficits Questionnaire - 5 item scale (PDQ-5) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-integrated tool (THINC-it) brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The cognitive questionnaire is called the Perceived Deficits Questionnaire - 5 item scale (PDQ-5). The questionnaire assesses self perceived cognition by asking questions about attention/concentration, retrospective memory, prospective memory, and planning/organization. Each item is rated on a 5-point scale ranging from 0 (never) to 5 (almost always). Higher scores indicate greater perceived deficits in cognition.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Choice Reaction Time | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The first objective cognitive test is called "spotter" and measures choice reaction time by calculating the total time that elapses between the presentation of a stimulus and the occurrence of a response in a task that requires a participant to make one of two different responses depending on which stimuli is presented. Less time between presentation of stimulus and occurrence of a response can be used as an indicator for better reaction time.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Working Memory | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The second objective cognitive test is called "Symbol Check" and is an n-back test. N-back tests measure working memory by presenting the subject with a sequence of stimuli, and the task consists of selecting the stimuli that was presented n steps earlier in the sequence. The greater amount of correct responses can be used as an indicator of better working memory.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Digit Symbol Substitution | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The third objective cognitive test is called "CodeBreaker" and is a Digit Symbol Substitution Test (DSST). DSST involves a key consisting of the numbers 1-6, each paired with a unique symbol. Below the key are a series of the numbers 1-6 in random order and repeated several times. Subjects must select the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured, with higher number of correct symbols indicating greater cognitive function.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Trail Making Test part B | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The fourth objective cognitive test is called "Trails" and is a version of the Trail Making Test part B (TMT-B). The subject is presented with numbers and letters in circles placed in random array on the screen. The subject must draw a line from one circle to the next in ascending order; however, s/he must alternate the circles with numbers in them and circles with letters in them (ie, 1-A-2-B-3-C etc). The TMT is a timed test and the goal is to complete the tests accurately and as quickly as possible. Less time to accurately complete the trial indicates greater cognitive function.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Implicit Suicidality | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Death Implicit Association Test (D-IAT) is a behavioral test that measures the strength of automatic (implicit) associations between concepts in people's minds relying on latency measures in a simple sorting task. The strength of an association between concepts of "death" and "ones self" is measured by the standardized mean difference score of the 'hypothesis-inconsistent' pairings and 'hypothesis-consistent' pairings
Changes in inflammatory markers | Participants will provide a blood sample prior to TMS treatment (baseline) and after TMS treatment (Week 4)
  Participants will provide blood samples to characterize inflammatory profiles. Human Cytokine Proinflammatory Focused 15-Plex Discovery Assay® Array (HDF15) will be used for quantification of proinflammatory cytokines in human blood plasma samples.
Change in functional Magnetic Resonance Imaging | MRI scan will be completed at baseline and week 4
  Change in resting state functional connectivity as determined by an fMRI.
Fibro vs Healthy Control functional Magnetic Resonance Imaging | MRI scan will be completed at baseline
  Baseline differences in functional activity and connectivity as determined by a fMRI acquisition between healthy controls and patients with fibromyalgia
Change in Magnetic Resonance (MR) spectroscopy | MRI scan will be completed at baseline and week 4
  Change in brain metabolites in regions of interest.
Fibro vs Healthy Control Magnetic Resonance (MR) spectroscopy | MRI scan will be completed at baseline
  Baseline differences in metabolites in regions of interest between healthy controls and patients with fibromyalgia
Neuromelanin | MRI scan will be completed at baseline
  Baseline differences in neuromelanin between healthy control and patients with fibromyalgia as measured by MRI
Quantitative Sensory Testing (QST) - Pain pressure thresholds via Algometry | QST will be completed at baseline and week 4
  Sensory perception will be assessed using a quantitative sensory testing battery. This will quantify multiple aspects of pain, including pain pressure thresholds using algometry. The pain pressure threshold is the point at which a non-painful pressure stimulus turns into a painful pressure sensation. Algometry will be administered at the trapezius and insertion point of the quadriceps. Subjects will be asked to indicate when the stimulus feels painful, which will terminate the application. The pressure will be measured as a range of 0 kPa-1,100 kPa. Higher values indicate higher pain threshold. This will be repeated 3 times at each site.
  Metrics from each of these tests will be compared between groups and overtime using ANCOVA models.
  In a separate set of analyses, the treatment end scores will be compared to healthy, matched control sample to determine treatment effects in relation to health. These will involve ANOVA or chi-square tests and Fisher's exact test where required
Quantitative Sensory Testing (QST) - Central sensitization via Temporal summation | QST will be completed at baseline and week 4
  Temporal summation will be used to measure central sensitization. Participants will be asked to rate the sensation of a weighted punctate probe (Range:0 "no pain" - 100 "worst pain imaginable") to a single stimulus and to a train of stimuli (10 identical stimuli repeated every second for 10 seconds). Central sensitization can be quantified by subtracting the rating of the single stimuli from the rating of the train of stimuli. Values greater than 0 indicate central sensitization, negative values will indicate a lack of central sensitization. This will be repeated 2 times (probes at force of 256mN and 512mN) at the non-dominant middle finger and patella.
  Metrics from each of these tests will be compared between groups and overtime using ANCOVA models.
  The treatment end scores will be compared to healthy, matched control sample to determine treatment effects in relation to health. These will involve ANOVA or chi-square tests and Fisher's exact test where required
Quantitative Sensory Testing (QST) - Conditioned pain modulation via cold-pressor conditioning | QST will be completed at baseline and week 4
  Sensory perception will be assessed using a quantitative sensory testing battery. This will quantify multiple aspects of pain, including cold-pressor conditioning to measure conditioned pain modulation, in which a hand is immersed in a 4-8°C water bath during pressure threshold testing of the opposite trapezius and compared to the baseline pain pressure threshold. The amount of pressure will be measured as a range of 0 kPa-1,100 kPa. Higher values indicate higher pain threshold. The time that the hand is in the water is approximately 30 seconds. This is repeated 3 times, with at least 2 minute breaks between each trial
  Metrics from each of these tests will be compared between groups and overtime using ANCOVA models.
  In a separate set of analyses, the treatment end scores will be compared to healthy, age-matched control sample to determine treatment effects in relation to health. These will involve ANOVA or chi-square tests and Fisher's exact test where required
Quantitative Sensory Testing (QST) - cold-pressor tolerance testing | QST will be completed at baseline and week 4
  Sensory perception will be assessed using a quantitative sensory testing battery. This will quantify multiple aspects of pain, cold pressor tolerance testing, in which a hand is placed in a 4-8°C water bath for 5 minutes, with numerical rating of level of discomfort every 30 seconds (Rating: 0 "no pain" - 100 "worst pain imaginable"). Participants may withdraw hand prior to 5 minutes if this becomes painful (rather than noxious).
  Time in cold water bath will also be indicative of cold pressor tolerance (more time indicating more cold tolerance).
  Metrics from each of these tests will be compared between groups and overtime using ANCOVA models.
  In a separate set of analyses, the treatment end scores will be compared to healthy, age-matched control sample to determine treatment effects in relation to health. These will involve ANOVA or chi-square tests and Fisher's exact test where required

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Daily Monday-Friday throughout study (4 weeks) and at one month follow up
  Adverse events will be tracked and recorded
Side Effects | The TSES will be administered at baseline, Week 2, Week 4, and at follow up (week 8)
  Side effects will be tracked through the Toronto Side Effects Scale (TSES). The TSES is a self reported questionnaire that assesses incidence, frequency, and severity of central nervous system, gastrointestinal, and sexual side effects. Individuals will be asked to rate frequency of each symptom within the last week on a 5-point scale, from "Never" (1) to "Everyday" (5). Severity of each symptom is similarly rated on a 5-point scale, from "No trouble" (1) to "Extreme Trouble" (5).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No